CLINICAL TRIAL: NCT06049511
Title: The Effect of the Oral Self-Care Protocol on Mucositis and Self-Care Agency According to Orem's Self-Care Deficiency Theory in Patients With Hematologic Malignancies Receiving High-Dose Chemotherapy: A Randomized Controlled Study
Brief Title: Oral Self Care Protocol and Oral Mucositis
Acronym: OSCP and OM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilek Eraslan, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Scientific Research Project
Record Dates: First submitted 2023-09-05; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Mucositis Oral
Keywords: oral mucositis; oral self care protocol; Orem's nursing theory; self-care agency
MeSH Terms: conditions — Stomatitis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: randomized controlled group
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The dentist who evaluated oral mucositis did not know which group the patients belonged to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): An oral self-care protocol, grounded in Orem's Self-Care Deficit theory and incorporating self-care behaviors, was implemented for the patients in the treatment group. The protocol consisted of several components, including the assessment of oral mucositis by the researcher and self-assessment of the oral cavity by the patients. It also involved oral care, teaching proper tooth brushing techniques, providing written materials, supplying an oral care kit, and offering patient and family education.
  Interventions: Behavioral: oral self care protocol
- control group (Other): The control group consisted of a total of 30 patients who met the selection criteria, willingly participated in the study, and were randomly assigned based on a predetermined randomization list. In the control group, the investigator did not administer any specific oral care intervention. Instead, the patients received standard nursing care provided at the clinic to prevent oral mucositis. Moreover, all patients in the control group were given the same mouthwashes (Benzydamine and Mycostatin) as those in the treatment group. However, the frequency and timing of oral care varied among the nurses in the clinic due to differences in work load and individual experience.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: oral self care protocol — An oral self-care protocol, grounded in Orem's Self-Care Deficit theory and incorporating self-care behaviors, was implemented for the patients in the treatment group. The protocol consisted of several components, including the assessment of oral mucositis by the researcher and self-assessment of the oral cavity by the patients. It also involved teaching proper tooth brushing techniques, providing written materials, supplying an oral care kit, and offering patient and family education. Interventions were made for 21 days from the beginning of chemotherapy treatment.
  Arms: intervention group
Behavioral: standard care — the patients received standard nursing care provided at the clinic to prevent oral mucositis.
  Arms: control group

SUMMARY:
Objective: This study was conducted in order to examine the effect of oral self-care protocol based on Orem's Self-Care Deficiency Theory on oral mucositis and self-care agency.

Method: This study was conducted as a randomized controlled trial between August 2021 and July 2022, patients with hematological malignancies receiving high-dose chemotherapy at the Izmir Ege University Faculty of Medicine Hospital and Izmir Training and Research Hospital. The sample of the study consisted of a total of 60 patients, including 30 application groups and 30 control groups, who met the inclusion criteria using the computer-based stratified randomization method. The study data were collected using "Patient Information Questionnaire," "WHO-Oral Mucositis Toxicity Scale," "Oral Assessment Guide," "Self-Care Agency Scale," "Data Collection Form Prepared According to Orem's Self-Care Deficiency Nursing Theory," "Oral Care Chart," and "Oral Cavity Photography." The oral self-care protocol, which includes training and oral care practices, was applied to the application group for 21 days from the beginning of chemotherapy treatment. The control group was not subjected to any oral care attempts by the researcher and received standard nursing care in the clinic. The data were evaluated by descriptive statistics, the Chi-square test, the Mann-Whitney U test, the Mc Ne-mar test, the Kappa compliance test, and the t test in dependent and independent groups. Keywords: chemotherapy; hematological malignancy; oral mucositis; oral self-care protocol; Orem's theory; self-care agency; nursing

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate,
* Have the ability to read and write,
* Volunteer for oral cavity photography,
* Possess a platelet value above 20,000/mm3, and
* Have intact oral mucous membrane integrity.

Exclusion Criteria:

* Who received combined radiotherapy and chemotherapy treatments
* Had incomplete questionnaire responses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
World Health Organization Oral Mucositis Toxicity Scale | 21 days
  to assess oral mucositis severity. The World Health Organization (WHO) classifies oral mucositis into different grades: grade 0 indicates no issues with the oral mucosa; grade 1 signifies mild local changes such as erythema and inflammation, with the ability to consume oral food; grade 2 involves mild pain, along with erythema, edema, inflammation, or ulcers, allowing unrestricted eating; grade 3 denotes painful erythema, edema, or ulcers without bleeding, necessitating a liquid food diet; and grade 4 represents extensive mucositis, severe pain, and bleeding, rendering oral feeding impossible.

SECONDARY OUTCOMES:
Oral assessment guide | 21 days
  assess their oral condition on a daily basis and serves as a valuable tool for monitoring the progression of mucositis and evaluating the effectiveness of treatment. This guide encompasses eight categories: voice, swallowing, lips, tongue, saliva, mucous membranes, gums, and teeth or dentures. Each category is assigned numerical values of 1, 2, or 3, representing normal findings (1 point) to severe findings (3 points). The cumulative score for all eight categories ranges from 8 points, indicating normal findings, to 24 points, denoting severe changes. A higher score indicates an increased risk of developing mucositis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Medical Faculty Hospital, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No